CLINICAL TRIAL: NCT06880653
Title: Examination of the Dose Response Relationship Between Physical Activity and Arthritis-Attributable Outcomes
Brief Title: Dose Response of Exercise for Arthritis Management
Acronym: DREAM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Christine A Pellegrini, PhD, Associate Professor, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00140006; U48DP006850 (NIH)
Record Dates: First submitted 2025-03-11; First posted 2025-03-18 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Arthritis; Rheumatoid Arthritis (RA); Gout; Fibromyalgia (FM); Osteoarthritis; Lupus Erythematosus, Systemic
Keywords: arthritis; exercise; physical activity
MeSH Terms: conditions — Arthritis; Arthritis, Rheumatoid; Gout; Fibromyalgia; Osteoarthritis; Lupus Erythematosus, Systemic; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 45 minutes/week (Experimental): Participants will be given a goal of 45 minutes/week of moderate-to-vigorous intensity physical activity
  Interventions: Behavioral: DREAM Adaptive Intervention
- 90 minutes/week (Experimental): Participants will be given a goal of 90 minutes/week of moderate-to-vigorous intensity physical activity
  Interventions: Behavioral: DREAM Adaptive Intervention
- 150 minutes/week (Experimental): Participants will be given a goal of 150 minutes/week of moderate-to-vigorous intensity physical activity
  Interventions: Behavioral: DREAM Adaptive Intervention

INTERVENTIONS:
Behavioral: DREAM Adaptive Intervention — 6-month physical activity program (Dose Response of Exercise for Arthritis Management (DREAM)) which includes monthly phone coaching, Walk With Ease Guidebook, behavioral lessons, and a Fitbit. Participants may receive additional contact (email, text, or phone) if they struggle to meet activity goal.

SUMMARY:
The purpose of the study is to see examine the effects of 3 different levels of physical activity (45 minutes/week, 90 minutes/week, or 150 minutes/week) on arthritis symptoms.

DETAILED DESCRIPTION:
All participants will be randomly assigned a physical activity goal (45 min/week, 90 min/week, or 150 min/week). To help participants achieve goals, they will receive a 6 month program which includes the Arthritis Foundation's Walk With Ease Guidebook, behavioral lessons, a Fitbit, and monthly coaching calls. Participants may also receive additional calls, texts, or emails if they are struggling to meet their physical activity goals.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Have a doctor diagnosed form of arthritis, rheumatoid arthritis, gout, lupus, or fibromyalgia
* Ability to read and write in English

Exclusion Criteria:

* Have any contraindications to exercise (besides arthritis)
* Engage in ≥30 min/week of Actigraph assessed MVPA
* Are pregnant, breastfeeding, or planning to become pregnant in the next year
* Are planning to relocate out of the Columbia, SC area in the next 12 months,
* Do not have a device compatible with Fitbit
* Have uncontrolled hypertension (e.g., systolic blood pressure > 160 mmHg or diastolic blood pressure > 100 mmHg)
* Plan to have a surgery that affects mobility in the next 12 months
* Have a serious cognitive impairment.
* Not willing to be randomized to any of the 3 conditions, do not believe they could adhere to the goals, or do not believe they could achieve the highest dose of activity (150 minutes/week).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 285 (Estimated)
Dates: Start 2025-03-28 (Actual); Primary Completion 2028-10-01 (Estimated); Study Completion 2029-04-30 (Estimated)

PRIMARY OUTCOMES:
Physical function (6 Minute Walk Test) | Baseline to 6 months
  Change in distance walked during the 6 minute walk test

SECONDARY OUTCOMES:
Physical function (6 Minute Walk Test) | Baseline to 12 months
  Change in distance walked during the 6 minute walk test
Physical function (chair stands) | Baseline to 6 months
  Change in chair stand repetitions
Physical function (chair stands) | Baseline to 12 months
  Change in chair stand repetitions
Health Related Quality of Life - Physical | Baseline to 6 months
  Change in the physical component score of the SF-12v2 Health Survey. Scores range from 0-100, with higher scores reflective of better health.
Health Related Quality of Life - Physical | Baseline to 12 months
  Change in the physical component score of the SF-12v2 Health Survey. Scores range from 0-100, with higher scores reflective of better health.
Health Related Quality of Life - Mental | Baseline to 6 months
  Change in the mental component score of the SF-12v2 Health Survey. Scores range from 0-100, with higher scores reflective of better health.
Health Related Quality of Life - Mental | Baseline to 12 months
  Change in the mental component score of the SF-12v2 Health Survey. Scores range from 0-100, with higher scores reflective of better health.
Pain intensity | Baseline to 6 months
  Change in pain as measured by a visual analog scale. Scores range from 0-100, with higher scores reflective of higher pain.
Pain intensity | Baseline to 12 months
  Change in pain as measured by a visual analog scale. Scores range from 0-100, with higher scores reflective of higher pain.
Depression symptoms | Baseline to 6 months
  Change in depression symptoms using the CES-D. Scores range from 0-60, with higher scores reflective of more depression symptoms.
Depression symptoms | Baseline to 12 months
  Change in depression symptoms using the CES-D. Change in depression symptoms using the CES-D. Scores range from 0-60, with higher scores reflective of more depression symptoms.

OTHER OUTCOMES:
Physical activity (min/week) | Baseline to 6 months
  Change in Actigraph-assessed moderate-to-vigorous intensity physical activity
Physical activity (min/week) | Baseline to 12 months
  Change in Actigraph-assessed moderate-to-vigorous intensity physical activity

CONTACTS AND LOCATIONS:
Overall Officials: Christine Pellegrini, PhD, Principal Investigator — University of South Carolina
Locations (1):
- University of South Carolina, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be made available within 30 months of the completion of the project.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: De-identified data will be made available within 30 months of the completion of the project.